CLINICAL TRIAL: NCT01634373
Title: An Open-Label, Randomised, 2-Period, 2-Treatment, 2-sequence, Crossover, Steady State Bioequivalence Study of Quetiapine Fumarate 300 mg Tablets [Test Formulation; Torrent Pharmaceuticals Ltd., India] Versus Seroquel® 300 mg Tablet [Reference Formulation; AstraZeneca, USA] in Schizophrenic Patients.
Brief Title: Steady State Bioequivalence Study of Torrent Pharmaceuticals Ltd's Bioequivalence Study of Torrent Pharmaceuticals Ltd's Quetiapine Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PK-08-111
Record Dates: First submitted 2012-06-27; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Torrent's Quetiapine Fumarate Tablets

SUMMARY:
Objective:

Primary objective was to study Steady-state bioequivalence of Torrent's Quetiapine Fumarate Tablets 300 mg.

Study Design:

Randomized, Two-Way, Crossover, multiple Dose, and Open-Label

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male of female
* Age: 25-65 years
* Patients who are receiving a stable daily dose of quetiapine 300 mg every 12 hourly for atlist one month
* Patient willing to adhere to the protocol requirements

Exclusion Criteria:

* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG.
* Significant orthostatic hypotension (i.e., a drop in systolic blood pressure of 30 mm Hg or more and/or a drop in diastolic blood pressure of 20 mm Hg or more on standing)
* Concurrent use of antihypertensive medication or any medication that might pre-dispose to orthostatic hypotension.
* History of allergic reactions to quetiapine or other chemically related psychotropic drugs.
* Concurrent primary psychiatric or neurological diagnosis including organic mental disorder, severe tardive dyskinesia, or idiopathic Parkinson's disease.
* Existence of any surgical or medical condition, which in the judgement of the Principal Investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of patients.
* Concurrent use of other drugs known to suppress bone marrow function.
* HIV, HCV, HBsAg positive.
* Expected changes in concomitant medications during the period of study.
* A history of epilepsy or risk for seizures
* positive urine drug of abuse test at enrollment.
* A history of alcohol or drug dependence by Diagnostic and statistical manual of Mental disorders IV(DSM-IV) criteria during the 6 month period immediately prior to study entry.
* A total white blood cell count below 4000/ml, or absolute neutrophil count below 2000/ml
* Female patients with pregnancy or Breast feeding or intend to become pregnant during the study and not able to follow contraception methods.
* History of multiple syncopal episodes.
* Administration any study drugs in last 3 months prior to entry in the study.
* History of significant blood loss due to any reason in the past 3 months.
* Any pre-existing bleeding disorder.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Asha Hospital, Hyderabad, India